CLINICAL TRIAL: NCT01194336
Title: Evaluation of Three Potential CNS Pretreatments for Soman Exposure - Huperzine A, Donepezil, and Galantamine - on Human Performance
Brief Title: Evaluation of Three Potential Central Nervous System (CNS) Pretreatments for Soman Exposure on Human Performance
Status: Completed | Type: Observational
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: WRAIR 1650; A-16072 (Other: HSRRB)
Record Dates: First submitted 2010-08-31; First posted 2010-09-03 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Biomarkers, Pharmacological
Keywords: Central nervous system; Cholinesterase; Neurocognitive performance testing
MeSH Terms: conditions — Butyrylcholinesterase deficiency | interventions — huperzine A; Donepezil; Galantamine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (7):
- Huperzine A: 100 ug
  Interventions: Drug: Huperzine A
- Huperzine A: 200 ug
  Interventions: Drug: Huperzine A
- Donepezil: 2.5 mg
  Interventions: Drug: Donepezil
- Donepezil: 5 mg
  Interventions: Drug: Donepezil
- Galantamine: 4 mg
  Interventions: Drug: Galantamine
- Galantamine: 8 mg
  Interventions: Drug: Galantamine
- Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Huperzine A — dosage form: tablet dose frequency: once only
  Groups: Huperzine A: 100 ug; Huperzine A: 200 ug
Drug: Donepezil — dosage form: tablet dosage frequency: once only
  Groups: Donepezil: 2.5 mg; Donepezil: 5 mg
Drug: Galantamine — dosage form: tablet dosage frequency: once only
  Groups: Galantamine: 4 mg; Galantamine: 8 mg
Other: Placebo — dosage form: tablet dosage frequency: once only
  Groups: Placebo

SUMMARY:
The primary objective of this study is to determine whether huperzine A, donepezil, and galantamine impact militarily relevant aspects of neurocognitive performance in humans, compared to placebo.

DETAILED DESCRIPTION:
The primary objective of this study is to determine whether huperzine A, donepezil, and galantamine impact militarily relevant aspects of neurocognitive performance in humans, compared to placebo.

Secondary: Secondary objectives are to correlate neurocognitive performance effects with degree of inhibition and therefore sequestration of red blood cell AChE by huperzine A, donepezil, and galantamine, and to monitor the safety of the study drugs in healthy adult (18-39 years) males and females.

In a double-blind, randomized, placebo-controlled, parallel-groups design, normal, healthy, adult male and female volunteers will be administered one of the drug/doses. They will be tested prior to and periodically for militarily relevant performance tasks for up to 8 hours post-dose and for cholinesterase levels via finger prick.

ELIGIBILITY:
Inclusion Criteria:

* All healthy men and women 18 to 39 years of age are eligible to participate.

Exclusion Criteria:

Must be able to swallow whole pills.

* Self-reported habitual nightly sleep amounts outside the target range of 6-8 hours (i.e., less than 6 hours per night or more than 8 hours per night, on average)
* Cardiovascular disease (to include but not limited to arrhythmias, valvular heart disease, congestive heart failure, family history of sudden cardiac death or myocardial infarction) as determined by participant self report.
* Current hypertension or high blood pressure (greater than 140/90)
* Neurologic disorder (to include but not limited to epilepsy or another seizure disorder, amnesia for any reason, hydrocephalus, MS, narcolepsy or other sleep disorders)
* Kidney disease
* History of psychiatric disorder requiring hospitalization or psychiatric medication for any length of time
* Beck Depression Inventory score of 14 or above
* Underlying pulmonary disease requiring daily inhaler use
* Regular nicotine use (or addiction) (defined as more than 1 cigarette or equivalent per week) within the last 3 years
* Heavy alcohol use (more than 2 drinks per day; http://www.cdc.gov/alcohol/faqs.htm#10)
* Use of other illicit drugs (to include but not limited to benzodiazepines, amphetamines, cocaine, marijuana)
* Known liver disease or liver abnormalities as determined by a laboratory test
* Known ulcer disease or risk of ulcer disease (stomach bleeding)
* Self-reported history of caffeine use in excess of 400 mg (8 caffeinated sodas or 3-4 cups, each ~ 6 oz, of coffee) per day on average
* Pregnancy (females)
* Breast-feeding (females)
* Prior anaphylactic reaction, angioedema, or other severe psychological reactions to any of the test compounds

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adults (18-39 years) males and females, military or civilian
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2012-02; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Observe military relevant neurocognitive performance in humans taking huperzine A, donepezil and galantamine compared to placebo. | 6pm Day 1 to 7pm Day 2
  The primary objective of this study is to determine whether huperzine A (a nutraceutical), donepezil (Aricept®), and galantamine (Razadyne®), impact militarily relevant aspects of neurocognitive performance in humans, compared to placebo.

SECONDARY OUTCOMES:
Correlate neurocognitive performance effects of huperzine A, donepezil and galantamine and to monitor the safety of the study drugs in healthy adults. | 6pm Day 1 to 7pm Day 2
  Secondary objectives are to correlate neurocognitive performance effects with degree of sequestration of red blood cell AChE by huperzine A, donepezil, and galantamine, and to monitor the safety of the study drugs in healthy adults.

CONTACTS AND LOCATIONS:
Overall Officials: MAJ James E Moon, MC, Principal Investigator — Walter Reed Army Institute of Research (WRAIR)
Locations (1):
- Walter Reed Army Institute of Research, Silver Spring, Maryland, United States